CLINICAL TRIAL: NCT03319277
Title: A Randomized-controlled Trial of Post-operative Opiate Quantities After Urogynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-1012
Record Dates: First submitted 2017-10-11; First posted 2017-10-24 (Actual); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Postoperative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine opiate prescription (Active Comparator): This arm will receive the standard post-discharge prescriptions of ibuprofen, docusate, acetaminophen, and polyethylene glycol. In addition, they will receive the standard amount of post-discharge opiate medications - 28 tablets of oxycodone 5mg.
  Interventions: Other: Routine opiate prescription
- Decreased opiate prescription (Experimental): This arm will receive the standard post-discharge prescriptions of ibuprofen, docusate, acetaminophen, and polyethylene glycol. In addition, they will receive the decreased amount of post-discharge opiate medications - 5 tablets of oxycodone 5mg with a paper prescription for an additional 10 tablets of oxycodone 5mg as a backup for uncontrolled pain.
  Interventions: Other: Decreased opiate prescription

INTERVENTIONS:
Other: Decreased opiate prescription — The experimental group will receive 5 tablets of oxycodone 5mg at time of discharge with a paper backup prescription for an additional 10 tablets.
  Arms: Decreased opiate prescription
Other: Routine opiate prescription — The comparator group will receive 28 tablets of oxycodone 5mg at time of discharge.
  Arms: Routine opiate prescription

SUMMARY:
This is a randomized controlled trial to determine the effect of decreased post-operative prescriptions of opiate medications after urogynecologic surgery.

DETAILED DESCRIPTION:
This is a randomized controlled trial to assess the hypothesis that patients prescribed fewer or no opiates will have no difference in satisfaction with pain control.

Safety/Data Monitoring:

Any adverse event or unanticipated events will be reported immediately to the IRB using IRB WebKit. All events will be recorded and kept in a research binder assigned to this study in a locked office. Monthly reviews during the study period will be done by all involved study staff members to ensure that events are not occurring, and if they are, that they are being handled and reported properly. The study will be terminated if over 50% of patients in the decreased opiate group request more or stronger medication during interim analysis or have >20% decreased satisfaction to the control group; this will be assessed monthly at the reviews mentioned above.

STUDY PROCEDURES Study Identification and Recruitment Potential subjects will be identified by members of the Center for Urogynecology and Pelvic Reconstructive Surgery at the Cleveland Clinic Main Campus. At the time of decision for surgery, attending staff who have been counseled about how to discuss the study will bring up the study. Fliers will be available to give to patients. Patients will be offered a visit with research staff at this time. They also will have the opportunity to meet research staff at their preop visit which is when consent forms would be signed and prescriptions given. Phone calls from research staff will also be made to interested patients or potential subjects. Eligible patients who agree to participate will be provided written informed consent administered by the collaborators listed on the IRB. Consents can be obtained at the Cleveland Clinic Main Campus or Fairview hospital.

Randomization All subjects will be scheduled for surgery by their surgeon. Consenting patients who meet inclusion criteria will be randomized into one of two arms: "routine opiate prescription" or "decreased opiate prescription" according to a computer-generated randomization schedule with random block sizes with the use of the JMP statistical software. The routine arm will receive twenty-eight tabs of oxycodone at discharge - thirty was the usual number prescribed for these surgeries, but new opiate prescribing guidelines limit the amount prescribed as 28 tablets based on morphine equivalent doses and a 7 day prescription limit. The decreased prescription arm will receive five tabs of oxycodone. All subjects will be instructed to use the opiate pills only as a back-up pain plan after the NSAID and acetaminophen. All subjects will be instructed to use the same schedule: schedule ibuprofen and acetaminophen for 3 days followed by these as needed. Subjects will have their prescriptions filled on day of discharge at the Cleveland Clinic pharmacy based on the randomization in addition to the following medications that per protocol all patients will receive unless contraindicated due to allergy/medication interaction: Colace (100mg tablets to take PO BID, #60), Miralax (17gm packets to take PO daily, #30), and ibuprofen (600mg tablets to take PO every 6 hours for 3 days postoperatively then as needed, #60. The use of scheduled NSAIDs is based on benefit of multimodal therapy in an effort to minimize opiate use. Despite these medications' potential effect to decrease effect seen between the study groups, their use in the trial provides increased clinical applicability.

Dispensing Medication If the patient approves to participate in the study, they will receive the allotted post-operative medication at time of discharge prescriptions for their postoperative medications as above at their preoperative visit. In addition, patients will also receive a sealed envelope with a prescription for a back-up supply of pain medication (10 pills of oxycodone 5mg). They will be instructed to fill these only if they run out of the previous supply and are still requiring stronger pain medication. Because of the way the prescription will be written (with instructions to the pharmacy not to fill before the date of post-operative day 2), they cannot automatically fill the same day as discharge (post-operative day 1) and this prescription is only valid for two weeks after this date. They will be instructed that if they require more pain medication than this, they will need to be seen. Patients will be provided with a daily pain and activity diary and medication log. At their 6-week postoperative visit, patients will bring in this diary as well as any remaining opiate medication and/or the sealed envelope containing the back-up prescription.

Data Collection & Management:

Other than the study forms, the electronic medical record (EPIC) will be used to obtain basic medical information including medical problems, height & weight/BMI, past surgeries, current medications, and allergies.

Preoperative data will include the following:

• Patient age, race and ethnicity, menopausal state, tobacco use, BMI, education level, patient income level

Peri-operative data will include the following:

* Surgery performed
* Surgical complications
* EBL (estimated blood loss)
* Hospital complications
* Delayed complications
* Prescribed medications (with detail given to agreement with randomization arm and if multimodal agents were not prescribed and for what reason)
* Post-operative pain scores at last RN assessment on day of discharge
* Medication records of quantity of narcotics used perioperatively (to be standardized to morphine equivalents)

Postoperative data will include the following:

* Patient's daily pain diaries including medications used which can be completed on paper diaries to be turned in at their post-operative visit OR entered electronically using REDCap (see below)
* Patient satisfaction with post-discharge pain control
* Patient's daily activities
* Whether patient received additional narcotic prescription through the following:

  * Study protocol through a phone call
  * Study protocol through an outpatient visit
  * Other (e.g. emergency room, urgent care)
* Patient satisfaction with bowel symptoms and constipation treatment as needed
* Number of pills used (as calculated by pill count or pain diary if pills not returned)
* Number of remaining pills (as calculated by pill count or pain diary if pills not returned)
* Patient's willingness to destroy remaining pills

Protection of each subject's personal health information will be a priority in this study. One master excel file containing subject personal information including name and medical record number will be kept in a password-protected file, on a designated protected research drive on a password-protected computer in a locked office at the Cleveland Clinic. In that file, each subject will be assigned a subject identification number that will be used for the purposes of data collection in order to de-identify subjects.

All paper forms used for data collection will be kept in a research cabinet dedicated to this project which will be locked at all times, in a locked office at the Cleveland Clinic. All forms will contain de-identified information - identification numbers will correspond to the subjects listed in the master excel file.

All study data will be transferred and managed electronically using REDCap (Research Electronic Data Capture). Each subject will be entered into REDCap using the assigned identification number from the master excel file. REDCap is a secure, web-based application designed to support data capture for research studies, providing user-friendly web-based case report forms, real-time data entry validation, audit trials, and a de-identified data export mechanism to common statistical packages. They system was developed by a multi-institutional consortium which was initiated at Vanderbilt University and includes the Cleveland Clinic. The database is hosted at the Cleveland Clinic Research Datacenter in the JJN basement and is managed by the Quantitative Health Sciences Department. The system is protected by a login and Secure Sockets Layers (SSL) encryption. Data collection is customized for each study based on a study-specific data dictionary defined by the research team with guidance from the REDCap administrator in Quantitative Health Sciences at the Cleveland Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or older
2. Women scheduled to undergo minimally invasive surgery within the urogynecology division at Cleveland Clinic with a plan to stay one night in the hospital afterwards for a benign indication which includes:

   * Vaginal hysterectomies with prolapse repair
   * Sacrospinous ligament fixations
   * Hysteropexy
   * Sacrocolpopexy
3. Women able to provide consent for research participation and to sign an informed consent

Exclusion Criteria:

* Women with chronic pain or chronic pain syndrome
* Women undergoing concurrent bowel surgery
* Women with pre-operative chronic opiate use
* Inability to comprehend written and/or spoken English
* Inability to provide informed consent
* Inability to take oxycodone
* Inability to take acetaminophen due to allergy or liver disease
* Women will be excluded if they undergo an unplanned laparotomy
* Pain catastrophization score

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily RW Davidson, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Routine Opiate Prescription | Decreased Opiate Prescription
Started | 59 | 59
Completed | 59 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Opiate Prescription | Decreased Opiate Prescription | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11.6) | 63 (9.0) | 62 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 56 | 106
  Black | 3 | 2 | 5
  Hispanic | 1 | 0 | 1
  Other | 3 | 1 | 4
  Unknown | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 59 | 118

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Adequate Satisfaction
Description: Patient satisfaction was easured by the way they answered the following question: "Overall, how satisfied are you with your pain medication at home since your surgery?" Their answers were recorded via a rated scale with five options: "Very Satisfied", "Somewhat Satisfied", "Neutral", "Somewhat Satisfied", and "Very Unsatisfied" which goes from most favorable to least favorable, respectively. Patients who answered either "Very Satisfied" or "Somewhat Satisfied" were defined a priori to have adequate satisfaction.
Time Frame: 6-weeks after surgery
Population: Two patients in the decreased opiate prescription group did not complete the follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Opiate Prescription | Decreased Opiate Prescription
Number analyzed (Participants) | 59 | 57
Participants | 55 | 53

2. Secondary Outcome: Number of Opiate Tablets Used by Patients
Description: Total number of prescribed tablets used by patients
Time Frame: 6-weeks after surgery
Measure: Median (Inter-Quartile Range); unit: number of tablets
Arm/Group | Routine Opiate Prescription | Decreased Opiate Prescription
Number analyzed (Participants) | 59 | 59
number of tablets | 3 [0 to 14] | 1 [0 to 3]

3. Secondary Outcome: Number of Patients Willing to Destroy Excess Remaining Opioid Tablets
Description: Patient answered "yes" to the following question: "Would you be willing to destroy any remaining opiate pain medication?"
Time Frame: 6-weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Opiate Prescription | Decreased Opiate Prescription
Number analyzed (Participants) | 53 | 53
Participants | 51 | 50

ADVERSE EVENTS:
Time Frame: 6-weeks after surgery
Arm/Group | Routine Opiate Prescription | Decreased Opiate Prescription
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT03319277/Prot_SAP_000.pdf